CLINICAL TRIAL: NCT05536947
Title: Micronutrient Bioavailability From Wheat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HR-18/19-5718
Record Dates: First submitted 2021-12-14; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard-milled Wholegrain (Active Comparator): Bread rolls prepared using standard-milled Wholegrain (75 g per bread roll, containing stable isotopes of Fe and Zn), with butter and strawberry jam.
  Interventions: Other: Bread product (standard milled)
- Micro-milled Wholegrain (Experimental): Bread rolls prepared using Micro-milled Wholegrain (75 g per bread roll, containing stable isotopes of Fe and Zn), with butter and strawberry jam.
  Interventions: Other: Bread Product (micro-milled)
- White flour fortified with standard milled Aleurone (Active Comparator): Bread rolls prepared using a white flour and standard-milled aleurone mix (75 g per bread roll, containing stable isotope of Fe), with butter and strawberry jam.
  Interventions: Other: Bread Product (standard aleurone)
- White flour fortified with micro-milled Aleurone (Experimental): Bread rolls prepared using a white flour and micro-milled aleurone mix (75 g per bread roll, containing stable isotope of Fe), with butter and strawberry jam.
  Interventions: Other: Bread product (micro-milled aleurone)

INTERVENTIONS:
Other: Bread product (standard milled) — Bread rolls made from standard milled flour.
  Arms: Standard-milled Wholegrain
Other: Bread Product (micro-milled) — Bread rolls made from micro-milled whole grain flour.
  Arms: Micro-milled Wholegrain
Other: Bread Product (standard aleurone) — Bread rolls made from white flour/standard milled aleurone mix
  Arms: White flour fortified with standard milled Aleurone
Other: Bread product (micro-milled aleurone) — Bread rolls made from white flour/micro-milled aleurone mix.
  Arms: White flour fortified with micro-milled Aleurone

SUMMARY:
The purpose of this study is to determine if physical disruption of wheat aleurone cell walls (micro-milling) increases micronutrient availability.

DETAILED DESCRIPTION:
This research project is a short-term dietary intervention study to investigate the bio-availability of iron and zinc from wheat. Approximately 50% of iron and 30% of zinc in the United Kingdom diet is provided by cereals and cereal products (e.g. bread and breakfast cereals). The localisation of both iron and zinc metals in wheat is largely confined to the aleurone layer, a single layer of cells located between the centre (endosperm) and outer layers (testa and pericarp). The aleurone layer is removed during the production of white flour. For this reason, since 1953 it has been mandatory to add iron to flours at the mill to restore iron to levels present in wholegrain flour (The Bread and Flour Regulations, 1998).

The investigators have shown that aleurone cells are resistant to physical disruption and digestion as they pass along the gastrointestinal tract and are excreted intact in faeces. The investigators believe that disruption of wheat aleurone cell walls prior to food manufacturing would therefore increase iron and zinc availability. Using wholegrain flour and purified wheat aleurone flour the investigators have shown that micro-milling, a process which reduces particle size of flour from approximately 100μm to 10μm, ruptures the aleurone cell walls, and increases iron availability, i.e. the amount absorbed by intestinal cells, compared with flour produced using standard milling techniques (which does not break down the aleurone layer).

Based on these initial findings, the current study therefore has 2 main aims:

(i) to determine whether physical disruption of the aleurone (by micro-milling) in wholegrain flour increases iron and zinc availability from wholegrain bread.

(ii) to determine whether addition of micro-milled aleurone flour to white flour increases iron availability from white bread.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menopausal women
* Serum ferritin below 30 μg/L
* Plasma zinc below 13.8 μmol/L.

Exclusion Criteria:

* Allergic to gluten or wheat
* Pregnant
* Post-menopausal women
* History of alcohol or substance abuse
* History of Cardiovascular Disease, diabetes, cancer, kidney, liver or intestinal disease, gastrointestinal disorder or use of drugs likely to alter gastrointestinal function.
* Donated blood recently (within 3 months prior to screening visit)
* Volunteers planning to take any mineral or vitamin supplements during the course of the study.

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Analysis of 57-Fe incorporation into erythrocytes | Through study completion, an average of 1 year
  Determines Fe incorporation from test meal into Red Blood Cells
Urinary excretion of Zinc | Through study completion, an average of 1 year
  Determine excretion of Zinc in urine samples to assess Zinc bioavailability

SECONDARY OUTCOMES:
Analysis of iron status biomarkers from blood samples | Through study completion, an average of 1 year
  Determine Hepcidin concentration from sample

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Sharp, PhD, Principal Investigator — King's College London, Department of Nutritional Sciences
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No